CLINICAL TRIAL: NCT00153569
Title: Phase II Study of Multiepitope Peptide Vaccination in Combination With Adjuvants GM-CSF and KLH in Metastatic Melanoma
Brief Title: Multiepitope Peptide Vaccination in Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HaemaCBFMM03
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2005-09

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Monophenol Monooxygenase; MAGEA3 protein, human

INTERVENTIONS:
Biological: Tyrosinase, MAGE-3, GnTV

SUMMARY:
This trial assesses the clinical efficacy of a multiepitope peptide vaccine with GM-CSF and KLH as immunological adjuvants in stage IV melanoma patients

ELIGIBILITY:
Inclusion Criteria:

* Metastatic melanoma
* HLA-A1, -A2, -A24, -B44

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2003-03; Study Completion 2005-09

PRIMARY OUTCOMES:
Clinical efficacy

SECONDARY OUTCOMES:
Immune response
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Keilholz, MD, Principal Investigator — Charité, CBF
Locations (1):
- Hem&Onc Charité CBF, Berlin, Germany

REFERENCES:
- [Background] Scheibenbogen C, Schadendorf D, Bechrakis NE, Nagorsen D, Hofmann U, Servetopoulou F, Letsch A, Philipp A, Foerster MH, Schmittel A, Thiel E, Keilholz U. Effects of granulocyte-macrophage colony-stimulating factor and foreign helper protein as immunologic adjuvants on the T-cell response to vaccination with tyrosinase peptides. Int J Cancer. 2003 Mar 20;104(2):188-94. doi: 10.1002/ijc.10961. PMID 12569574